CLINICAL TRIAL: NCT01827332
Title: Effect of Oxytocin on Craving and Therapy Response in Marijuana-dependent Individuals
Brief Title: Effect of Oxytocin on Craving and Therapy Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Aimee McRae-Clark, Associate Professor of Psychiatry, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20991
Record Dates: First submitted 2013-04-02; First posted 2013-04-09 (Estimated); Results first posted 2016-11-11 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Marijuana Dependence
Keywords: marijuana; substance abuse; drug abuse; marijuana dependence; drug addiction
MeSH Terms: conditions — Marijuana Abuse; Substance-Related Disorders | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Active Comparator): intranasal administration
  Interventions: Drug: Oxytocin
- Saline (Placebo Comparator): intranasal administration
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Oxytocin — Subjects will be administered 40 IUs of oxytocin nasal spray or matching placebo prior to two individual sessions of MET.
  Other Names: Pitocin
  Arms: Oxytocin
Drug: Saline — Subjects will be administered 40 IUs of oxytocin nasal spray or matching placebo prior to two individual sessions of MET.
  Other Names: Placebo
  Arms: Saline

SUMMARY:
The purpose of this study is to examine the impact of a medication called oxytocin on marijuana use and therapy response in people who frequently use marijuana.

DETAILED DESCRIPTION:
Oxytocin has been shown to promote trust, social bonding, and calmness; however, its potential additive effects with a therapy intervention have not been explored in marijuana-dependent individuals. In the proposed study, the impact of intranasal oxytocin on therapy effectiveness and marijuana use outcomes following a brief therapy intervention will be investigated. It is hypothesized that oxytocin administration (vs. placebo) will improve treatment satisfaction and decrease marijuana use.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
2. Subjects must meet DSM-IV criteria for current marijuana dependence (within the past three months). While individuals may also meet criteria for abuse of other substances, they must identify marijuana as their primary substance of abuse and must not meet criteria for dependence on any other substance (except nicotine) within the last 60 days.
3. Subjects must consent to remain abstinent from alcohol for 24 hours and other drugs of abuse (except nicotine and marijuana) for three days immediately prior to study procedures. Subjects must abstain from marijuana for 24 hours prior to testing. By restricting marijuana use as proposed, subjects should not be under the acute effects of marijuana.
4. Subjects must consent to random assignment.

Exclusion Criteria:

1. Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control.
2. Subjects with evidence of or a history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal, or neurological disease including diabetes, as these conditions may affect physiological/subjective responses.
3. Subjects with a history of or current psychotic disorder or bipolar affective disorder as these may interfere with subjective measurements.
4. Subjects who pose a current suicidal or homicidal risk.
5. Subjects taking any psychotropic medications, including SRI's or other antidepressants, opiates or opiate antagonists because these may affect test response. Individuals who take stimulants for treatment of ADHD will be allowed to participate.
6. Subjects with any acute illness or fever. Individuals who otherwise meet study criteria will be rescheduled for evaluation for participation.
7. Subjects who are unwilling or unable to maintain abstinence from alcohol and marijuana for 24 hours and other drugs of abuse (except nicotine) for three days prior to study procedures.
8. Subjects meeting DSM-IV criteria for substance dependence (other than nicotine or marijuana) within the past 60 days.
9. Subjects who, in the investigator's opinion, would be unable to comply with study procedures or assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee L McRae-Clark, PharmD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited between July 2014 and May 2015 primarily through media and internet advertisements.
Groups:
- Oxytocin: intranasal administration
  Oxytocin: Subjects will be administered 40 IUs of oxytocin nasal spray prior to two individual sessions of MET.
- Saline: intranasal administration
  Saline: Subjects will be administered 40 IUs of saline nasal spray (placebo) prior to two individual sessions of MET.
Period: Overall Study
Arm/Group | Oxytocin | Saline
Started | 8 | 8
Completed | 6 | 7
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Saline | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Therapy Session Satisfaction (as Measured by Subjective Report)
Description: After MET sessions, subjects completed the Session Rating Scale (SRS, Miller et al). This visual analog scale is comprised of 4 items for which participants rate their therapy experience in terms of relationship, goals and topics, approach/method, and overall, with minimum score 0 representing most dissatisfied and maximum score 10 representing most satisfied. Outcome measure reported below represents SRS score at last MET session.
Time Frame: Within 5 minutes of completing a 45-60 minute Motivational Enhancement Therapy (MET) session at last session visit
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Oxytocin | Saline
Number analyzed (Participants) | 6 | 7
units on a scale | 9.8 (0.4) | 9.7 (0.3)

2. Secondary Outcome: Marijuana Use (as Measured by Subjective Report of Number of Daily Smoking Sessions )
Description: Subjects' marijuana use was measured via self-report of number of smoking sessions per day (Time Line Followback). The average number of daily sessions were calculated per group, with data presented below representing the change in amount of daily smoking sessions per group from first MET session to last MET session.
Time Frame: Self-report of average daily smoking sessions at MET Session 1 and last MET session 3
Measure: Mean (Standard Error); unit: daily smoking sessions
Arm/Group | Oxytocin | Saline
Number analyzed (Participants) | 6 | 7
daily smoking sessions | -1.39 (0.42) | -0.22 (0.44)

ADVERSE EVENTS:
Arm/Group | Oxytocin | Saline
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=8) | Saline (N=8)
Headache (General disorders) | 0 (0) | 2 (2)
Other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations included small sample size and limited generalizability as individuals with other substance use disorders were excluded from participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No